CLINICAL TRIAL: NCT06100822
Title: Managing Chronic Tendon Pain by Repurposing Metformin
Brief Title: Managing Chronic Tendon Pain by Metformin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: James Wang (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, James Wang, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY23040151; HT9425-23-1-0712 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2023-10-09; First posted 2023-10-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Tendinopathy; Chronic Pain; Achilles Tendinopathy
Keywords: Achilles Tendon; Metformin; Achilles Tendinopathy; Chronic Pain
MeSH Terms: conditions — Tendinopathy; Chronic Pain | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Group, Placebo Capsules (Placebo Comparator): Placebo Group (n=20) Week 1: One placebo capsule (500 mg) daily Week 2: Two placebo capsules (1,000 mg) daily Week 3: Three placebo capsules (1,500 mg) daily Week 4-16: Four placebo capsules (2,000 mg) daily
  Interventions: Drug: Placebo
- Treatment Group, Metformin Capsules (Experimental): Treatment Group (n=20) Week 1: One metformin ER capsule (500 mg) daily Week 2: Two metformin (ER) capsules (1,000 mg) daily Week 3: Three metformin (ER) capsules (1,500 mg) daily Week 4-16: Four metformin (ER) capsules (2,000 mg) daily
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 500 mg capsules of Metformin Extended Release
  Other Names: Glucophage; Glucophage XR; Metformin Extended Release; Metformin ER
  Arms: Treatment Group, Metformin Capsules
Drug: Placebo — 500 mg capsules of placebo pills
  Arms: Placebo Group, Placebo Capsules

SUMMARY:
The purpose of the current exploratory clinical trial is to determine the effect of oral ingestion of metformin (OIM) in non-diabetic patients with chronic Achilles tendon pain. The trial has two aims; 1) to assess the effects of OIM treatment on tendon pain, and 2) to determine the effects of OIM capsules on tendon healing and repair. Twenty participants will be treated with metformin capsules for 16 weeks combined with a home exercise program. A comparison group of 20 participants will be treated with placebo tablets along with home exercise program.

DETAILED DESCRIPTION:
This is a blinded and randomized controlled trial that focuses on the treatment effects of metformin (Met) on chronic tendon pain, healing, and repair in midportion Achilles tendinopathy. We will include a total 40 patients randomly divided into two equal groups:

Group 1: Home Exercise Program + Placebo as a control group

Group 2: Home Exercise Program + Oral Ingestion of Metformin

Patients in group 1 will receive placebo capsules,1 capsule (500 mg) daily for week one, 2 capsules (1,000 mg) daily for week two, 3 capsules daily for week 3 (1,500 mg), and 4 capsules daily (2,000 mg) for weeks 4-16. Patients in group 2 will receive metformin capsules,1 capsule (500 mg) daily for week one, 2 capsules (1,000 mg) daily for week two, 3 capsules daily for week 3 (1,500 mg), and 4 capsules daily (2,000 mg) for weeks 4-16. All patients will participate in a home exercise program through MedBridge, a HIPAA-compliant participant portal currently used by physical therapists at University of Pittsburgh Medical Center. There are 3 visits for this study. Visits include a Screening/Baseline visit, week 4 and week 16 visit. During each visit, participants will answer questions, complete functional testing, and undergo an ultrasound of the Achilles Tendon.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent for participation
* Clinical diagnosis of Achilles tendinopathy
* Pain disability index score of between 20 - 70 points (0-100 scale VISA-A)
* Sonopalpation tenderness with tendon thickening and/or loss of fibrillary architecture.
* Ability to read, speak, and understand English

Exclusion Criteria:

* Any intervention (corticosteroids or other orthobiologic intervention as injection) to targeted tissue within the last 6 months.
* Previous Achilles tendon surgery.
* Known platelet abnormality or hematological disorder.
* Presence of other conditions that might affect the functional scale of the indexed limb.
* Unwillingness to be randomized.
* Body Mass Index (BMI) greater than 30.
* Occult tear in the indexed tendon.
* Systemic inflammatory disease.
* Use of fluoroquinolone in the past 6 months.
* Subjects must not be pregnant or breastfeeding, or planning to become pregnant or breastfeed during the course of the trial
* Chronic kidney disease (eGFR <60)
* Diagnosis of diabetes mellitus or elevated HbA1c at screening (> 6.5)
* Unable to take an oral medication in a non crushable pill form
* Taking metformin presently or within the last 6 months
* History of allergy to metformin
* History of lactic acidosis or elevated lactate at screening (> 2.2)
* Severe Hepatic dysfunction
* Currently taking a diabetic medication such as sitagliptin, saxagliptin, linagliptin, alogliptin, sitagliptin with metformin
* Currently taking a Carbonic anhydrase inhibitor such as topiramate, zonisamide, acetazolamide, dichlorphenamide, methazolamide
* Currently taking cimetidine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Victorian Institute of Sport Assessment - Achilles (VISA-A) Score | baseline, 4 weeks, 16 weeks
  The VISA-A is a self-administered questionnaire that asks about Achilles tendon pain, function, and activity. Scores range from 0 to 100 with a low score indicating more severe pain.

SECONDARY OUTCOMES:
Change in VAS score | baseline, 4 weeks, 16 weeks
  The VAS is a self-administered questionnaire that asks about pain. Scores range from 0 to 10 with a high score indicating more severe pain.
Change in tendon thickness | baseline, 4 weeks, 16 weeks
  Images of the Achilles tendon in long axis will be acquired using B-mode ultrasound imaging. Maximum Achilles tendon thickness (mm) will be measured by a blinded investigator.
Change in tendon cross-sectional area | baseline, 4 weeks, 16 weeks
  Images of the Achilles tendon in short axis will be acquired using B-mode ultrasound imaging. Maximum Achilles tendon cross-sectional area (mm^2) will be measured by a blinded investigator.
Change in tendon neovascularization | baseline, 4 weeks, 16 weeks
  Achilles tendon neovascularization will be evaluated using the 5-point modified Ohberg scale:
  0 - no vessels visible
  1. one vessel, mostly anterior to the tendon
  2. one or two vessels throughout the tendon
  3. three vessels throughout the tendon
  4. more than three vessels throughout the tendon
Change in tendon hypoechogenicity | baseline, 4 weeks, 16 weeks
  Hypoechogenicity is indicative of disruption of the normal fibrillar structure of the Achilles tendon. Achilles tendon hypoechogenicity will be evaluated using a semi-quantitative 3-point scale:
  0 - no hypoechogenicity
  1. - Heterogeneous echotexture with diffuse hypoechogenicity between fibrillar echoes and/or foci of discontinuity in collagen fibrillar echoes
  2. - Heterogeneous echotexture with discrete hypoechoic area/s of >1mm and/or presence of intrasubstance tears
Change in maximum number of heel raises | baseline, 4 weeks, 16 weeks
  The subject will stand barefoot on a 10° incline board and perform heel raises at a rate of 30 Hz (2 seconds per repetition, pace provided by audible metronome), while keeping their knee straight. Subjects will be allowed to have 2 fingertips per hand at shoulder height against the wall for balance. Participants will stop when they are unable to perform any additional repetitions, or if they fail to maintain proper form. Number of repetitions will be recorded.
Change in heel raise height | baseline, 4 weeks, 16 weeks
  The subject will stand barefoot on a 10° incline board and perform heel raises at a rate of 30 Hz (2 seconds per repetition, pace provided by audible metronome), while keeping their knee straight. Subjects will be allowed to have 2 fingertips per hand at shoulder height against the wall for balance. Participants will stop when they are unable to perform any additional repetitions, or if they fail to maintain proper form. Maximum height of heel rise achieved during repetitions will be measured using the Calf Raise App.
Change in heel raise work | baseline, 4 weeks, 16 weeks
  The subject will stand barefoot on a 10° incline board and perform heel raises at a rate of 30 Hz (2 seconds per repetition, pace provided by audible metronome), while keeping their knee straight. Subjects will be allowed to have 2 fingertips per hand at shoulder height against the wall for balance. Participants will stop when they are unable to perform any additional repetitions, or if they fail to maintain proper form. Total work (body weight x total distance) will be measured using the Calf Raise App.
Change in counter movement jump height | baseline, 4 weeks, 16 weeks
  Subjects will stand on a single leg with their hands behind their back, bend their knee as much as desired, and jump as high as possible from flat ground. Three trials will be performed. Jump height will be determined using the My Jump2 App and the highest jump height will be utilized in further analysis.
Change in drop counter movement jump height | baseline, 4 weeks, 16 weeks
  Subjects will stand on a single leg on top of an 8" plyometric box, with their hands behind their back. They will be asked to "fall" down to the floor and then immediately jump as high as possible from flat ground. Three trials will be performed. Jump height will be analyzed using the My Jump2 App and the highest jump height will be utilized in further analysis.
Change in VAS score during hopping | baseline, 4 weeks, 16 weeks
  Subjects will be asked to complete two 2 trials of 25 single leg hops at a natural cadence similar to jumping rope (~2 jumps/second). Subjects will be asked to rate their pain during the exercise using VAS (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: James H Wang, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement. For more information or to submit a request, please contact wanghc@pitt.edu